CLINICAL TRIAL: NCT02139371
Title: 64Cu-DOTA-AE105. Evaluation of a New Radiotracer Targeting uPAR (Urokinase Plasminogen Activator Receptor) for Positron Emission Tomography Imaging of the Invasive Cancer Phenotype. First in Man.
Brief Title: Evaluation of a New Radiotracer (64Cu-DOTA-AE105) for Diagnosing Aggressive Cancer With Positron Emission Tomography
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Dorthe Skovgaard, MD, Phd, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-574
Record Dates: First submitted 2014-05-12; First posted 2014-05-15 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Breast Cancer; Prostate Cancer; Urinary Bladder Cancer
Keywords: Positron Emission Tomography; Uroplasminogen Plasminogen Activator Receptor; Breast cancer; Prostate cancer; Urinary bladder cancer; Biodistribution; Radiation exposure
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 64Cu-DOTA-AE105 PET (Experimental): One injection of 64-Cu-DOTA-AE105 (app. 200 Mbq IV) followed by 3 PET scans 1,3 and 24 hours post injection
  Interventions: Other: Injection of 64Cu-DOTA-AE105

INTERVENTIONS:
Other: Injection of 64Cu-DOTA-AE105 — One injection of 64Cu-DOTA-AE105 (app. 200 Mbq) followed by Positron Emission Tomography Scan 1, 3 and 24 hours post injection

SUMMARY:
The primary objective of the study is to test a new radiotracer called 64Cu-DOTA-AE105 for PET imaging of uPAR (urokinase plasminogen activator receptor). The tracer has the potential of identifying the invasive cancer phenotype, thereby distinguishing between aggressive and less aggressive tumors. This is a first in human study to test the radiotracer in cancer patients. The biodistribution and tumor uptake will be evaluated by repeated PET imaging (1,3 and 24 hours post injection).

DETAILED DESCRIPTION:
The primary objective of the study is to test a new radiotracer called 64Cu-DOTA-AE105 for PET imaging of uPAR (urokinase plasminogen activator receptor). The tracer has the potential of identifying the invasive cancer phenotype, thereby distinguishing between aggressive and less aggressive tumors. This is a first in human study to test the radiotracer in cancer patients. The biodistribution and tumor uptake will be evaluated by repeated PET imaging (1,3 and 24 hours post injection). The primary end points are Biodistribution and dosimetry of 64Cu-DOTA-AE105. In addition, the quantitative uptake of 64Cu-DOTA-AE105 in tumors and expression of uPAR in tumor tissue obtained by surgery or biopsies (either 14 days before (only biopsies) or after the PET scans) will be compared to validate the image-derived data on UPAR expression

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of cancer of prostate, breast or urinary bladder
* capable of understanding and giving full informed consent

Exclusion Criteria:

* pregnancy
* lactation
* contraindication for the use of intravenous CT contrast-agencies
* claustrophobia
* other current/or former diagnosed cancers, except non melanoma skin cancer or carcinoma in situ cervicis uteri

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Biodistribution | 24 hours
  The patients will be PET scanned 1, 3 and 24 hours post injection of the radiotracer 64Cu-DOTA-AE105. These different timepoints will be used for assessment of biodistribution
Dosimetry | 24 hours
  The patients will be PET scanned 1, 3 and 24 hours post injection of the radiotracer 64Cu-DOTA-AE105. These different timepoints will be used for calculation of dosimetry

SECONDARY OUTCOMES:
Expression of UPAR in tumor tissue | 24 hours
  Tumor uptake of 64Cu-DOTA-AE105 will be compared with expression of uPAR (using immunohistochemistry and ELISA) in tumor tissue obtained from biopsies/or operative removal of the tumors.
Quantitative uptake of UPAR in tumor tissue | 24 hours
  The patients will be PET scanned 1, 3 and 24 hours post injection of the radiotracer 64Cu-DOTA-AE105. These different timepoints will be used for assessment of tumor uptake of 64Cu-DOTA-AE105 will be assessed by PET scans 1, 3 and 24 hours post injection

CONTACTS AND LOCATIONS:
Overall Officials: Dorthe Skovgaard, MD, Phd, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Clinical Physiology, Nuclear Medicine and PET, Rigshospitalet, Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Background] Persson M, Madsen J, Ostergaard S, Jensen MM, Jorgensen JT, Juhl K, Lehmann C, Ploug M, Kjaer A. Quantitative PET of human urokinase-type plasminogen activator receptor with 64Cu-DOTA-AE105: implications for visualizing cancer invasion. J Nucl Med. 2012 Jan;53(1):138-45. doi: 10.2967/jnumed.110.083386. PMID 22213823